CLINICAL TRIAL: NCT01913834
Title: A Single-centre, Open-label, Five-way Crossover Study in Healthy Female Participants to Assess the Pharmacokinetics of Nasally Administered Formulations of Teriparatide Compared to a Subcutaneous Injection.
Brief Title: Nasally and sc Administered Teriparatide in Healthy Volunteers
Acronym: NINTTO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13MP002; Grant Ref: EP/K502364/1 (Other Grant/Funding Number: TSB CR&D)
Record Dates: First submitted 2013-06-26; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Osteoporosis
Keywords: Parathyroid hormone 1-34
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Forsteo (Active Comparator): Synthetic PTH 1-34 Single dose Subcutaneous administration 20.0 micrograms
  Interventions: Drug: Forsteo
- CP046 PTH CriticalSorb 22.5 R (Experimental): Synthetic PTH 1-34 Single dose Nasal administration rexam device 22.5 micrograms
  Interventions: Drug: CP046 PTH CriticalSorb
- CP046 PTH CriticalSorb 45.0 R (Experimental): Synthetic PTH 1-34 Single dose Nasal administration rexam device 45.0 micrograms
  Interventions: Drug: CP046 PTH CriticalSorb
- CP046 PTH CriticalSorb 90.0 R (Experimental): Synthetic PTH 1-34 Single dose Nasal administration rexam device 90.0 micrograms
  Interventions: Drug: CP046 PTH CriticalSorb
- CP046 PTH CriticalSorb 90.0 O (Experimental): Synthetic PTH 1-34 Single dose Nasal administration 90 micrograms
  Interventions: Drug: CP046 PTH CriticalSorb

INTERVENTIONS:
Drug: Forsteo — Subcutaneous administration 20 micrograms
  Other Names: teriparatide
  Arms: Forsteo
Drug: CP046 PTH CriticalSorb — Comparison of different doses of drug and nasal delivery devices
  Other Names: teriparatide
  Arms: CP046 PTH CriticalSorb 22.5 R; CP046 PTH CriticalSorb 45.0 R; CP046 PTH CriticalSorb 90.0 O; CP046 PTH CriticalSorb 90.0 R

SUMMARY:
Osteoporosis is a reduction in bone density that increases the risk of fractures; particularly of the spine, hip and wrist. Osteoporosis is estimated to affect 200 million women worldwide - approximately one tenth of women aged 60, one-fifth of women aged 70, two-fifths of women aged 80 and two-thirds of women aged 90. Treating osteoporosis and the associated fractures costs the NHS more than two billion pounds per annum.

Teriparatide is a drug currently prescribed for some osteoporosis patients by their doctor to be taken by injection. It is currently the only drug available which promotes the deposition of new bone as opposed to preventing resorption. This is the drug treatment we will be studying in this clinical trial.

The drug is of a type that cannot normally be taken as a swallowed pill. This type of drugs tends to be delivered by injection, as is currently the case for teriparatide. Injections have numerous limitations and are disliked by patients.

This trial will assess how well the nasal spray devices work, how long the drug stays in the nose and also how well the drug enters the bloodstream.

DETAILED DESCRIPTION:
This study aims to look at how teriparatide spreads through the nose and into the blood stream when it is given as a liquid with a nasal delivery system called CriticalSorb™. CriticalSorb has been developed by Critical Pharmaceuticals to improve the absorption of drugs through the nose into the blood stream in the hope that it will replace injections. For part of the study a radioactive compound (routinely used in the nuclear medicine clinic for diagnosis) will be added to the formulation in order to investigate how the formulation spreads through nose after it is sprayed.

The study is being carried out in postmenopausal females aged greater than 55 years of age as osteoporosis commonly affects these women. The study will involve 8 visits.

The first visit will be to assess eligibility. On visit 2 the participants will receive an injection of the teriparatide. On visits 2-6 the participants will receive a nasal dose of teriparatide via nasal devices at different dose levels, blood samples will be taken to measure drug levels following dosing.

For visits 5 and 6 the nasal dose will have a radioactive marker added and gamma camera imaging will also be carried out. These visits will also compare two different nasal devices.

Visit 7 will be a follow up visit. There will be one further visit during the study to acquire a MRI scan of the head that will assist analysis of the scintigraphic images.

ELIGIBILITY:
Inclusion Criteria:

* Be a postmenopausal healthy female and aged greater than 55 years of age
* Be able to give voluntary informed consent and from whom written consent to participate has been obtained
* Be able to understand the study, willing to co-operate with the study procedures and able to attend all study assessments
* Be willing to abstain from alcohol for 24 hours before each dose and until the end of each study day
* Be willing to abstain from smoking for 24 hours before each dose and until the end of each study day
* Be willing to avoid caffeine from midnight the evening prior to each study day

Exclusion Criteria:

* Have a history of alcohol or drug abuse and failure of urine tests for drug abuse
* Have had any investigational drug administered within the previous 3 months.
* Failed to satisfy the investigator's assessment of fitness to participate based on a completed health screening
* Have consumed alcohol or tobacco within 24 hours of start of each study day
* Have consumed caffeinated drink after midnight prior to each study day
* Have participated in a similar study involving the use of radioisotopes in the previous 3 months such that participating in the current study would exceed the recommended yearly exposure limit (5mSv)
* Have any presently active infectious diseases (such as influenza)
* Have a known hypersensitivity to teriparatide or to any of the excipients in the formulation
* Have a history of nasal disorders/problems
* Have a history of allergic rhinitis
* Have an increased baseline risk of osteosarcoma
* Have Paget's disease
* Have a history of any malignancy or radiotherapy
* Have a history of diabetes
* Have a history of hypercalcaemia
* Are taking any forbidden medications - see Appendix 2
* Inability to use both of the intranasal delivery devices
* Have a condition that prohibits MRI scans
* Have positive HIV or Hepatitis B or C test results or engage in a lifestyle that increases the risk of the possibility of these infections

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve (AUC) of teriparatide for six hours after each single administration. | predose, 0,1,2,3,4,6, hours post-dose
Peak plasma concentration (cmax) of teriparatide for six hours after each single administration. | predose, 0,1,2,3,4,6 hours post-dose

SECONDARY OUTCOMES:
The percentage of radiolabelled formultation deposited and cleared from the nose measured by gamma scintigraphy | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tahir Masud, MRCP, FRCP, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom